CLINICAL TRIAL: NCT03735901
Title: Enhancement of Stroke Rehabilitation With Levodopa (ESTREL): a Randomized Placebo-controlled Trial
Brief Title: Enhancement of Stroke Rehabilitation With Levodopa
Acronym: ESTREL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-02021; me16Engelter
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Acute Stroke; Stroke Rehabilitation
Keywords: Levodopa / Carbidopa; Fugl-Meyer-Motor-Assessment (FMMA); Acute ischemic stroke; Acute hemorrhagic stroke; Rehabilitation; Recovery; Randomized controlled trial
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Carbidopa

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized 1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention (Active Comparator): White Investigational Medicinal Product (IMP)- capsules of a combination of IMP Levodopa 100mg/Carbidopa 25mg.
  Interventions: Drug: IMP Levodopa 100mg/Carbidopa 25mg
- Control Intervention (Placebo Comparator): Matching placebo, identical in aspect, texture, and taste when compared to the IMP. Procedures regarding route of administration, study treatment duration and treatment phases will be identical in the IMP- and the placebo-group.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: IMP Levodopa 100mg/Carbidopa 25mg — Study treatment will comprise 3 phases:
  1. Dose escalation phase: On day 1-3, patients will receive IMP solely in the morning; on day 4-6 in the morning and at lunch time;
  2. full study treatment phase: from day 7 to day 34, 3 times per day (tid).
  3. Treatment will stop with a tapering phase: On day 35-37, patients will receive IMP in the morning and at lunch time; on day 38 and 39 solely in the morning.
  Arms: Experimental Intervention
Drug: Matching placebo — Study treatment will comprise 3 phases:
  1. Dose escalation phase: On day 1-3, patients will receive Placebo solely in the morning; on day 4-6 in the morning and at lunch time;
  2. full study treatment phase: from day 7 to day 34, Placebo capsules 3 times per day (tid).
  3. Treatment will stop with a tapering phase: On day 35-37, patients will receive Placebo in the morning and at lunch time; on day 38 and 39 solely in the morning.
  Arms: Control Intervention

SUMMARY:
Trial investigates the benefits and harms of Levodopa /Carbidopa 100/25mg compared to placebo (given in addition to standardized rehabilitation based on the principles of motor learning) and whether there is an association with a patient-relevant enhancement of functional recovery in acute stroke patients. Study participants will be randomized 1:1.

DETAILED DESCRIPTION:
Trial investigates whether Levodopa/Carbidopa compared to placebo given in addition to standardized rehabilitative therapy in patients with acute stroke is associated with

a) patient relevant improvements of physical function b) improvement in patient-self assessed general health aspects, pain, mood, anxiety, fatigue and social participation c) long-term sustainability of a patient-relevant improvement of motor function d) improvement of selective hand and wrist movement e) a higher rate of patients walking independently of the help of another person.

f) less severe impairment g) a higher level of activity of daily living h) improvements of quality of life (i) better cognitive performance (j) no signals of harms (i.e. indications for increased all-cause mortality, recurrent stroke, serious adverse events, and non-serious, pre-specified adverse events possibly related to the IMP)

Estrel-Longterm: optional prolongation of the observational study phase. To investigate the long-term outcomes of our study population the investigator aim to offer an optional prolongation of the observational phase to the participants through regular structured (once yearly) telephone visits.

The telephone visits will be carried out annually for the following 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic or hemorrhagic (i.e. intracerebral hemorrhage excluding subarachnoid hemorrhage and cerebral venous sinus thrombosis) stroke ≤ 7 days prior to randomization
* Clinically meaningful hemiparesis (i.e. scoring a total of ≥ 3 points on the following NIH stroke scale score items (i) motor arm, (ii) motor leg, (iii) limb ataxia; a distal arm paresis is equivalent to one of the aforementioned (i-iii))
* Time of randomization ≥24-hours since thrombolysis or thrombectomy
* In-hospital rehabilitation required
* Capable to participate in standardized rehabilitation therapy
* Informed consent of patient or next of kin

Exclusion Criteria:

* Diagnosis of Parkinson's Disease
* Use of Levodopa mandatory according to judgement of treating physician
* Inability or unwillingness to comply with study procedures including adherence to study drug intake (orally, or via nasogastric tube or percutaneous endoscopic gastrostomy tube)
* Severe aphasia (i.e. unable to follow two-stage-commands)
* Previously dependent in the basal activities of daily living (defined as modified Ranking Scale prior to stroke > 3)
* Pre-existing hemiparesis
* Known hypersensitivity to Levodopa/Carbidopa and other contraindications for Levodopa/Carbidopa as outlined in the summary of product characteristics
* Women who are pregnant or breast feeding, or who intend to become pregnant during the course of the study. Women of childbearing age must take a pregnancy test to be eligible for the study.
* Lack of safe contraception, defined as: Female Participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the Investigator in individual cases. Female Participants who are surgically sterilized / hysterectomized or post- menopausal for longer than 2 years are not considered as being of child- bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer-Motor Assessment Score (FMMA) | Assessed 3 months +/- 14 days after randomization
  FMMA is a stroke-specific impairment index designed to assess motor recovery. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale (0=cannot perform; 1=performs partially and 2= performs fully). FMMA total scores range from 0 (no movements) to 100 (normal movements) with 66 points for movements of the upper limbs (FMMA-UE) and 34 for those of the lower limbs (FMMA-LE). A difference of 5.25 points for the upper extremity and 6 points for the lower extremity part of the score are described as minimal clinically important difference. For this study, based on these data, 6 points difference are considered a patient-relevant difference between both treatment groups for the primary endpoint.

SECONDARY OUTCOMES:
NIH-Stroke Scale Score (NIHSS) | Assessed at Day 0 (Randomization), 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12 months +/- 30 days after randomization
  To objectively quantify the impairment caused by a stroke. NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For this study, an extra item for distal arm paresis was included (score from 0-2). For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42 (+4 for distal arm paresis), with the minimum score being a 0.
Modified Rankin Scale Score (mRS) | Assessed at Day 0 (Randomization), 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12/24/36/48/60 months +/- 30 days after randomization
  Scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Stroke rehabilitation outcomes for disease specific morbidity and quality of life - PROMIS 29 | Assessed 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12 months +/- 30 days after randomization
  Patient-self-assessment in the following categories: 1) physical function, 2) anxiety, 3) depression, 4) fatigue, 5) sleep disturbance, 6) ability to participate in social roles and activities, 7) pain interference and 8) pain intensity. Each of the domains 1 to 7 are assessed with 4 questions. Items are scored on 1 of 5 levels based on the ability of the participant to perform activities or the self-assessment of the participant in the various domains. Pain intensity is scored on a visual analogue scale of 0 to 10.
Stroke rehabilitation outcomes for disease specific morbidity and quality of life - PROMIS 10 | Assessed 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12/24/36/48/60 months +/- 30 days after randomization
  Patient-self-assessment Patient-Reported Outcomes Measurement Information System (PROMIS) 10 addresses general health aspects, quality of life, pain, mood, anxiety, fatigue and social participation; PROMIS-10 covers the outcome domains considered most important
Patient-reported assessment of relevance of motor improvement | Assessed 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12/24/36/48/60 months +/- 30 days after randomization
  Patients Questionnaire asking whether there is improvement in motor function since the last study visit and if so, whether this improvement is relevant in patients' personal perception (yes/ no).
Rivermead Mobility Index (RMI) | Assessed at Day 0 (Randomization), 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12/24/36/48/60 months +/- 30 days after randomization
  15 items that measure the ability of patients to make postural adjustments (e.g, move in bed), transfer (e.g. between bed to chair), walk, and use stairs and is scored from 0-15 Points. A RMI score of ≥ 7 translates into the ability of the patient walking independently of the assistance of another Person.
Mortality (of any cause) | Throughout the whole study period from Day 1 to Visit 12/24/36/48/60 months +/- 30 days after randomization
  death rate
Recurrent stroke (any type) | Throughout the whole study period from Day 1 to Visit 12/24/36/48/60 months +/- 30 days after randomization
  recurrent stroke (any type)
Pre- specified Adverse Events of Interest | Throughout the study period from Day 1 to Visit 3 ( 3 months +/- 14 days after randomization)
  Nausea, Vomiting, Taste disturbances, Dry mouth, Anorexia, Arrhythmias, Postural hypotension Syncope (unconsciousness for a short time as a result of reduced blood flow to the brain), drowsiness (including sudden onset of sleep) Fatigue, Dementia, Psychoses (a distorted perception of reality), Hallucinations, Confusion, Euphoria, Abnormal dreams, Insomnia, Depression, Anxiety, Dizziness, Dystonia (involuntary contractions), Dyskinesia (inability to control voluntary movements), Chorea (sudden twitching of the face and shoulders)
Motricity Index (MI) | Assessed at Day 0 (Randomization), 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12 months +/- 30 days after randomization
  Two subscales, one for the upper extremity (UE) (total score range 0 to 100) and one for the lower extremity (LE) (total score range 0 to 100). It measures isometric muscle strength (0 = no movement; 100 = normal)
Trunk Control Test (TCT) | Assessed at Day 0 (Randomization), 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12 months +/- 30 days after randomization
  Assesses the trunk abilities of the patient , contains 4 items, with item scores ranging from 0 to 25. The sitting balance item assesses the patients' ability to sit during 30 seconds without trunk and feet support and has a predictive value for recovery of walking poststroke
Action Research Arm Test (ARAT) | Assessed at Day 0 (Randomization), 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12 months +/- 30 days after randomization
  Assesses the patients' ability to grasp (subscale with 6 items), grip (subscale with 4 items), pinch (subscale with 6 items) and perform gross movements (subscale with 3 items) with the upper extremity. Score: 0 = no movement / 1= movement task is partially performed / 2 = movement task is completed but takes abnormally long / 3 = movement is performed normally
Box- and Block Test (BBT) | Assessed at Day 0 (Randomization), 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12 months +/- 30 days after randomization
  Patients (seated in front of a square box with two compartments) are asked to move as many wooden cubes as possible from one compartment to the other within 60 seconds of testing time.
Functional Ambulation Categories (FAC) | Assessed at Day 0 (Randomization), 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12/24/36/48/60 months +/- 30 days after randomization
  Classification (score range 0 to 5) regarding the ability to walk independently, with or without a walking aid and takes the type of walking surface into account.
  Rating:
  0 = Patient cannot walk, or needs help from 2 or more persons
  1. = Patient needs firm continuous support from 1 person who helps carrying weight and with balance
  2. = Patient needs continuous or intermittent support of one person to help with balance and coordination
  3. = Patient requires verbal supervision or stand-by help from one person without physical contact
  4. = Patient can walk independently on level ground, but requires help on stairs, slopes or uneven surfaces
  5. = Patient can walk independently anywhere
Ten-Meter Walk Test (10MWT) | Assessed at Day 0 (Randomization), 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12 months +/- 30 days after randomization
  Walking speed and cadence over a 10 meter track at both a comfortable and a maximum Speed; time in seconds over 10-meter walking distance
Jamar dynamometer testing (JDT) | Assessed at Day 0 (Randomization), 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12 months +/- 30 days after randomization
  grip strength and strength of the forearm (in kilogram)
Montreal Cognitive Assessment (MoCA) | Assessed at Day 0 (Randomization), 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12 months +/- 30 days after randomization
  Assesses cognitive domains: Short-term memory recall task (5 points).Visuospatial abilities assessed using clock-drawing task (3 points) and 3-dimensional cube copy (1 point). Executive functions assessed using alternation task. Attention, concentration, working memory evaluated using a sustained attention task (target detection using tapping; 1 point), serial subtraction task (3 points), digits forward and backward (1 point each). Languages assessed using 3-item confrontation naming task with low-familiarity animals (lion, camel, rhinoceros; 3 points), repetition of 2 complex sentences (2 points), and fluency task. Orientation to time and place evaluated by asking for date and city in which the test is occurring (6 points). A score of 26 or over is considered to be normal (range 0 to 30)
Daily activity measurement with movement sensor | Assessed at Day 0 (Randomization), 5 weeks after randomization, 3 months +/- 14 days after randomization, 6 months +/- 20 days after randomization and 12 months +/- 30 days after randomization
  Movement sensors allow assessment of physical activity engagement and upper limb use in daily life situations without physically hampering the patient in the performance of their daily activities
Serious Adverse Event (SAE) | Throughout the study period from Day 1 to Visit 3 ( 3 months +/- 14 days after randomization)
  Any untoward medical occurrence that:
  * results in death,
  * is life-threatening,
  * requires in-patient hospitalization or prolongation of existing hospitalisation,
  * results in persistent or significant disability/incapacity, or
  * is a congenital anomaly/birth defect
Fugl-Meyer-Motor Assessment Score (FMMA) | Assessed at Day 0 (Randomization), 5 weeks after randomization, 6 months +/- 20 days after randomization and 12 months +/- 30 days after randomization
  FMMA is a stroke-specific impairment index designed to assess motor recovery. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale (0=cannot perform; 1=performs partially and 2= performs fully). FMMA total scores range from 0 (no movements) to 100 (normal movements) with 66 points for movements of the upper limbs (FMMA-UE) and 34 for those of the lower limbs (FMMA-LE). A difference of 5.25 points for the upper extremity and 6 points for the lower extremity part of the score are described as minimal clinically important difference. For this study, based on these data, 6 points difference are considered a patient-relevant difference between both treatment groups for the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Engelter, Prof. MD, Principal Investigator — Felix-Platter Spital Basel
Locations (24):
- Switzerland (24):
  - Kantonsspital Aarau, Neurozentrum, Aarau
  - RehaClinic AG, Bad Zurzach
  - Kantonsspital Baden, Baden
  - Felix Platter Spital, Basel
  - Stroke-Center Universitätsspital Basel, Basel
  - Inselspital, Universitätsklinik für Neurologie, Bern
  - Kantonsspital Graubünden, Departement Innere Medizin / Neurologie, Chur
  - HFR Fribourg Hopital Cantonal, U. de Neurologie, Fribourg
  - Centre hospitalier universitaire vaudois, Service de Neurologie, Lausanne
  - HFR Meyriez-Murten, Clinique de Réhabilitation, Meyriez
  - Kantonsspital Münsterlingen, Münsterlingen
  - Reha Rheinfelden, Rheinfelden
  - Kantonsspital St.Gallen, Klinik für Neurologie, Sankt Gallen
  - Hôpital du Valais - Sion, Service de neurologie, Sion
  - Hôpital du Valais - Sion, Sion
  - Rehazentrum Valens, Klinik für Neurologie und Neurorehabilitation, Valens
  - Cereneo Schweiz AG, Vitznau
  - Zürcher RehaZentrum Wald, Wald
  - Rheinburg Klinik AG, Walzenhausen
  - Kantonsspital Winterthur, Winterthur
  - Rehaklinik Zihlschlacht, Zihlschlacht
  - Klinik Lengg AG, Zurich
  - Head Stroke Center Klinik Hirslanden, Zurich
  - Universitätsspital Zürich, Klinik für Neurologie, Zurich

REFERENCES:
- [Derived] Engelter ST, Kaufmann JE, Zietz A, Luft AR, Polymeris A, Altersberger VL, Wiesner K, Wiegert M, Held JPO, Rottenberger Y, Schwarz A, Medlin F, Accolla EA, Foucras S, Kagi G, De Marchis GM, Politz S, Greulich M, Tarnutzer AA, Sturzenegger R, Katan M, Fischer U, Nedeltchev K, Schar J, Van Den Keybus Deglon K, Rapin PA, Salerno A, Seiffge DJ, Auer E, Lippert J, Bonati LH, Schuster-Amft C, Gaumann S, Chabwine JN, Humm A, Moller JC, Schweinfurther R, Bujan B, Jedrysiak P, Sandor PS, Gonzenbach R, Mylius V, Lutz D, Lienert C, Peters N, Michel P, Muri RM, Schadelin S, Hemkens LG, Ford GA, Lyrer PA, Gensicke H, Traenka C; ESTREL Investigators. Levodopa Added to Stroke Rehabilitation: The ESTREL Randomized Clinical Trial. JAMA. 2025 Nov 4;334(17):1523-1532. doi: 10.1001/jama.2025.15185. PMID 40982270